CLINICAL TRIAL: NCT01694927
Title: Autologous Mesenchymal Stem Cells in Spinal Cord Injury (SCI) Patients
Acronym: MSC-SCI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Clínica Las Condes. LIT INNOVA CORFO (Other)
Responsible Party: Sponsor-Investigator, Clínica Las Condes. LIT INNOVA CORFO, Clinical Researcher LIT. Innova CORFO 09IEI6568, Clinica las Condes, Chile
Organization: Clinica las Condes, Chile (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIT-2012-ACF-001
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Spinal Cord Injury
Keywords: Mesenchymal stem cell; Spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mesenchymal Stem cells (Experimental)
  Interventions: Procedure: Autologous Mesenchymal Stem Cells

INTERVENTIONS:
Procedure: Autologous Mesenchymal Stem Cells — Expanded Intralesional Autologous Mesenchymal Stem Cells Transplantation

SUMMARY:
The aim of this study is to evaluate the use of autologous expanded mesenchymal stem cells intralesional transplantation as a safe and potentially beneficial treatment for patients with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* American Spinal Injury Association Impairment (ASIA) Scale A, B and C
* Cervical (under C4), thoracic o lumbar spine lesion
* Complete or Incomplete SCI
* Platelet count over 100.000/ul

Exclusion Criteria:

* Acute SCI (less than 3 months)
* Active infectious diseases
* Pregnancy
* Neurodegenerative diseases
* Primary hematologic diseases
* Coagulopathies
* Hepatic dysfunction
* Pregnancy

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Safety of Autologous Expanded Mesenchymal Stem Cells transplantation in SCI patients | 3 months

SECONDARY OUTCOMES:
Functional improvement in muscle strength | 1 year
  According to motor index score
Functional Improvement in sphincters control | 1 year
Functional improvement in spasticity control | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Chahín, MD, Principal Investigator — Clínica Las Condes, Santiago; Rodrigo M Mardones, MD, Study Director — Clínica Las Condes, Santiago; Catalina Larrain, MD, Study Chair — Clínica Las Condes, Santiago
Locations (1):
- Clínica Las Condes, Santiago, RM, Chile

REFERENCES:
- [Result] Pal R, Venkataramana NK, Bansal A, Balaraju S, Jan M, Chandra R, Dixit A, Rauthan A, Murgod U, Totey S. Ex vivo-expanded autologous bone marrow-derived mesenchymal stromal cells in human spinal cord injury/paraplegia: a pilot clinical study. Cytotherapy. 2009;11(7):897-911. doi: 10.3109/14653240903253857. PMID 19903102
- [Result] Ra JC, Shin IS, Kim SH, Kang SK, Kang BC, Lee HY, Kim YJ, Jo JY, Yoon EJ, Choi HJ, Kwon E. Safety of intravenous infusion of human adipose tissue-derived mesenchymal stem cells in animals and humans. Stem Cells Dev. 2011 Aug;20(8):1297-308. doi: 10.1089/scd.2010.0466. Epub 2011 Mar 17. PMID 21303266
- [Result] Moviglia GA, Fernandez Vina R, Brizuela JA, Saslavsky J, Vrsalovic F, Varela G, Bastos F, Farina P, Etchegaray G, Barbieri M, Martinez G, Picasso F, Schmidt Y, Brizuela P, Gaeta CA, Costanzo H, Moviglia Brandolino MT, Merino S, Pes ME, Veloso MJ, Rugilo C, Tamer I, Shuster GS. Combined protocol of cell therapy for chronic spinal cord injury. Report on the electrical and functional recovery of two patients. Cytotherapy. 2006;8(3):202-9. doi: 10.1080/14653240600736048. PMID 16793729